CLINICAL TRIAL: NCT04366973
Title: New Care Pathways to Achieve HCV Elimination in the Community: Real-world Outcomes From HCV Infected Patients Treated in Addiction Centers in France
Brief Title: A Study Describing the Care Cascade and Effectiveness and Safety of Glecaprevir/Pibrentasvir in Adult Participants With Hepatitis C Virus in French Addiction Centers
Acronym: NeoVie
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-127
Record Dates: First submitted 2020-04-28; First posted 2020-04-29 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: Hepatitis C Virus; HCV; glecaprevir/pibrentasvir; Maviret
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with Hepatitis C Virus With or Without Treatment: This study includes 3 populations for analysis:
  Target Population (TP): Defined as all participants enrolled in the study regardless of whether treated for HCV or not.
  Core Population (CP): Defined as all participants of the TP who have been prescribed glecaprevir/pibrentasvir (G/P) and started treatment.
  Safety Population (SP): Defined as all participants who received at least one dose of G/P.

SUMMARY:
Hepatitis C Virus is liver disease and is a leading cause of death and morbidity with around 71 million people affected worldwide. Widespread availability of highly effective direct-acting antivirals (DAAs) have dramatically changed the treatment landscape of HCV with a cure rate of over 95%. In May 2019, French Health Authorities expanded prescription abilities to all physicians treating adult treatment-naive patients with HCV without cirrhosis of the liver. This study will assess the treatment uptake and barriers to treatment by non-HCV specialist in France in community-based addiction centers. Beyond these evaluations, data on health resource utilization in addiction centers, level of knowledge of both patients and providers on HCV infection and treatment, care cascade, effectiveness and safety of Glecaprevir/Pibrentasvir among patients treated in addiction centers and evolution of addiction behavior after treatment are of specific interest.

Glecaprevir/Pibrentasvir is a drug approved to treat HCV. About 400 Adult participants with a confirmed positive HCV ribonucleic acid (RNA) test will be enrolled in the study at approximately 30 addiction centers in France.

All participants will attend an inclusion visit. Participants who are not prescribed Glecaprevir/Pibrentasvir at the inclusion visit will have no further follow-up in the study. Participants who are prescribed Glecaprevir/Pibrentasvir will take three tablets once daily. The duration of the study is approximately 12 months.

All study visits will occur during routine clinical practice but there may be a higher burden for participants prescribed Glecaprevir/Pibrentasvir. These participants will be asked to complete questionnaires after each visit.

ELIGIBILITY:
Inclusion Criteria:

* Followed in an addiction center.
* Confirmed positive for HCV ribonucleic acid (RNA).

Exclusion Criteria:

-None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants treated with glecaprevir/pibrentasvir for confirmed positive Hepatitis C Virus.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with and without Hepatitis C Virus (HCV) treatment prescribed at end of the inclusion visit. | Inclusion visit (Week 0)
  Percentage of participants with and without HCV treatment prescribed at end of the inclusion visit. Criteria for treatment choice and reasons for treatment refusal will be described.

SECONDARY OUTCOMES:
Health Care Resources and Utilization | Inclusion visit (Week 0)
  HCRU in the addiction centers will be described on the basis of declarative questionnaires completed at time of the study implementation (yearly number of people followed, health resources, staffing, formation of center team, capabilities regarding HCV screening, specialized consultations in hepatology, and liver fibrosis tests).
Level of HCV infection knowledge | Inclusion visit (Week 0)
  The level of knowledge of both patients and providers on HCV infection will be described on the basis of declarative questionnaires. For patients, analysis will be performed in the TP population and according to patient subgroups (with and without HCV treatment).
Determinants associated with initiation of HCV treatment | Inclusion visit (Week 0)
  Criteria for treatment choice or no treatment uptake assessed by physician, patient, and disease characteristics.
Data and disease characteristics from patients with and without HCV treatment | Inclusion visit (Week 0)
  Data and disease characteristics from patients with and without HCV treatment.
Number of participants with HCV Antibodies (HCV Ab) | Inclusion visit (Week 0)
  Number of participants with HCV Antibodies (HCV Ab).
Number of participants with HCV RNA | Inclusion visit (Week 0)
  Number of participants with HCV RNA.
Time from HCV Ab to HCV RNA | Inclusion visit (Week 0)
  Time from HCV Ab to HCV RNA.
Time from HCV RNA to end of treatment | Approximately 12 months
  Time from HCV RNA to end of treatment.
Number of participants who completed treatment | Approximately 12 months
  Number of participants who completed treatment.
Percentage of participants achieving SVR12 | Approximately 12 months
  SVR12 defined as HCV RNA under the lower limit of quantification (LLOQ) 12 weeks after the last dose of treatment with a sensitive polymerase chain reaction (PCR) test.
Percentage of cured participants willing to share their experience with other substance abuse patients. | Approximately 12 months
  Percentage of cured participants willing to share their experience with other substance abuse patients at the SVR12 visit and up to 6 months after the SVR12 visit.
Number of participants achieving sustained viral response at 12 weeks (SVR12) | Approximately 12 months
  Number of participants achieving sustained viral response at 12 weeks (SVR12).
Time to SVR12 | Approximately 12 months
  Time to SVR12
Number of people in charge of patient follow-up | Approximately 12 months
  Number of people in charge of patient follow-up including physicians, nurses, social workers.
Percentage of participants with treatment adherence | Approximately 12 months
  Defined as the percentage of participants who have taken the target dose according to participant reporting.
Patient Reported Quality of Life | Approximately 12 months
  Anxiety and depression questionnaires and global assessment using visual analog scale.
Number of participants with addictive behaviors | Approximately 12 months
  Addictive behaviors of participants (alcohol and drug consumption) will be assessed by participant-completed questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (30):
- France (30):
  - Centre de soin d'accompagnement et de prevention en addictologie- CHU Archet 2 /ID# 218682, Nice, Alpes-Maritimes
  - Centre de Soins d'Accompagnement et de Prevention en Addictologie-Tempo Oppelia /ID# 218701, Valence, Drome
  - CSAPA Bagnols sur ceze /ID# 233397, Bagnols-sur-Cèze, Gard
  - Centre de soin d'accompagnement et de prevention en addictologie- L'ENVOL /ID# 218680, Nîmes, Gard
  - CEID Bordeaux /ID# 221517, Bordeaux, Gironde
  - Centre de Soins d'Accompagnement et de Prevention en Addictologie- Arc en ciel /ID# 218700, Montpellier, Herault
  - Centre de soin d'accompagnement et prevention en addictologie-UTTD Montpellier /ID# 218683, Montpellier, Herault
  - Csapa Doaur Nevez de Ploermel /Id# 240583, Ploërmel, Morbihan
  - Centres de Soin d'Accompagnement et de Prevention en Addictologie-Les WADS CMSEA /ID# 218671, Metz, Moselle
  - Centre de Soins Accompagnement et de Prevention en Addictologie-Boris Vian /ID# 221284, Lille, Nord
  - Association Tremplin 17 - Saintes /ID# 218708, Saintes, Nouvelle-Aquitaine
  - Centre de soins d'accompagnement et de prevention en addictologie-ANPAA 82 /ID# 218675, Montauban, Occitanie
  - Centre Hospitalier Le Vinatier - Service universitaire d'addictologie de Lyon /ID# 218695, Bron, Rhone
  - Centre de Soins Accompagnement et de Prevention en Addictologie-Antibes /ID# 221277, Antibes
  - Centres de Soin d'Accompagnement et de Prevention en Addictologie -Bayonne /ID# 218673, Bayonne
  - CHU Clermont Ferrand - Hopital Gabriel Montpied /ID# 221278, Clermont-Ferrand
  - Centre de Soins Accompagnement et de Prevention en Addictologie - AGORA /ID# 223793, Cognac
  - Centre de Soins Accompagnement et de Prevention en Addictologie - ARGILE /ID# 223792, Colmar
  - Centre de Soins d'Accompagnement et de Prevention en Addictologie-ANPAA 21 /ID# 222909, Fontaine-lès-Dijon
  - Centre de Soins Accompagnement et de Prevention en Addictologie-CICAT /ID# 221281, Le Coudray
  - Centre Bobillot - Limoges /ID# 221922, Limoges
  - Centre de Soins d'Accompagnement et de Prevention en Addictologie- Le Sémaphore /ID# 222954, Marseille
  - Centre de Soins d'Accompagnement et de Prevention en Addictologie- Le Cap /ID# 222776, Mulhouse
  - Clinique Jules Verne /ID# 241666, Nantes
  - Centre de Soins d'Accompagnement et de Prevention en Addictologie- Malaussena /ID# 218703, Nice
  - Centre de Soins d'Accompagnement et de Prevention en Addictologie-Nova Dona /ID# 221516, Paris
  - CSAPA CAARUD Aurore EGO /ID# 225050, Paris
  - CEID Bearn addictions /ID# 221279, Pau
  - Centre de soin d'accompagnement et de prevention en addictologie -ITHAQUE /ID# 218678, Strasbourg
  - Centre de soin d'accompagnement et de prevention en addictologie-Paul Guiraud /ID# 218710, Bagneux, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.rxabbvie.com/